CLINICAL TRIAL: NCT07263204
Title: Precision Diagnosis and Prognostic Prediction of Hypertrophic Cardiomyopathy Using Artificial Intelligence: A Multicenter Study
Brief Title: AI-Enabled Diagnosis and Prognosis of Hypertrophic Cardiomyopathy
Status: Recruiting | Type: Observational
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Other Study IDs: 2024-1546
Record Dates: First submitted 2025-11-17; First posted 2025-12-04 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-01

CONDITIONS: Hypertrophic Cardiomyopathy (HCM); Left Ventricular Hypertrophy
MeSH Terms: conditions — Cardiomyopathy, Hypertrophic; Hypertrophy, Left Ventricular

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- HCM: diagnosed with hypertrophic cardiomyopathy by echocardiography and cardiac magnetic resonance imaging
- phenocopy: patients with left-ventricular hypertrophy attributable to non-hypertrophic cardiomyopathy conditions
- normal control: healthy individuals without myocardial hypertrophy

SUMMARY:
By harnessing artificial intelligence to decode the 12-lead electrocardiogram, the project will enable precise ECG-based phenotyping of hypertrophic cardiomyopathy-accurately classifying septal, apical, and other morphologic subtypes-while simultaneously differentiating HCM from hypertensive heart disease, aortic stenosis, and other phenocopy disorders.

DETAILED DESCRIPTION:
To overcome the twin bottlenecks of late detection and poor inter-centre reproducibility, the project leverages a large, multicentre historical cohort and anchors its pipeline on the 12-lead ECG-an inexpensive, ubiquitously available signal that can be captured in any department. Using deep-learning architectures augmented with attention mechanisms, we will develop (1) a discriminative model that separates HCM from phenocopies and normal hearts, and (2) an algorithmic framework that remains stable across devices and populations. Model governance will be embedded through version-controlled releases, cloud-edge deployment, and an "offline replay" evaluation loop, producing an end-to-end evidence chain that mirrors real-world clinical workflows.

ELIGIBILITY:
Inclusion Criteria:

1. Adults aged ≥ 18 years.
2. HCM cohort: Adults diagnosed with hypertrophic cardiomyopathy in accordance with the *2023 Chinese Guidelines for the Diagnosis and Treatment of Hypertrophic Cardiomyopathy in Adults*.
3. HCM phenocopy cohort: Adults with an LV wall thickness ≥ 13 mm at any site on echocardiography.
4. Healthy-control cohort: Adults with no history of cardiac disease and no evidence of myocardial hypertrophy on echocardiography.

Exclusion Criteria:

Patients from whom analyzable ECG data cannot be obtained.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 1. HCM cohort: Adults diagnosed with hypertrophic cardiomyopathy in accordance with the *2023 Chinese Guidelines for the Diagnosis and Treatment of Hypertrophic Cardiomyopathy in Adults*.
  2. HCM phenocopy cohort: Adults with an LV wall thickness ≥ 13 mm at any site on echocardiography.
  3. Healthy-control cohort: Adults with no history of cardiac disease and no evidence of myocardial hypertrophy on echocardiography.
Sampling Method: Non-Probability Sample
Enrollment: 15000 (Estimated)
Dates: Start 2025-01-01 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
model diagnostic performance | year 2
  Model performance was evaluated using calculated metrics including accuracy, sensitivity, specificity, and the area under the ROC curve (AUC).

SECONDARY OUTCOMES:
model diagnostic performance | year 2
  The accuracy rate of the model's phenotype-specific classification for patients with different patterns of myocardial hypertrophy
the model's generalizability | year 2
  The model's diagnostic performance on the external, multicentre validation cohort, including overall accuracy, sensitivity, specificity, and area under the ROC curve (AUC).

CONTACTS AND LOCATIONS:
Locations (1):
- Second Affiliated Hospital, Zhejiang University School of Medicine, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No